CLINICAL TRIAL: NCT04692285
Title: Targeting New Receptors in Dystonia: Electrophysiological and Neuroimaging Correlates of the Effect of Zolpidem, a Selective Agonist of Benzodiazepine Subtype Receptor alfa1, in Different Forms of Primary Focal Dystonia
Brief Title: Electrophysiological and Neuroimaging Correlates of the Effect of Zolpidem in Patients With Focal Dystonia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Medical Centre Ljubljana (Other)
Collaborators: Slovenian Research Agency (Other); Clinical Centre of Serbia (Other)
Responsible Party: Principal Investigator, Maja Kojović, doc. dr. Maja Kojović, dr. med., University Medical Centre Ljubljana
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 0120-232/2016
Record Dates: First submitted 2020-12-23; First posted 2020-12-31 (Actual); Last update posted 2023-12-04 (Actual); Status verified 2023-11

CONDITIONS: Focal Dystonia
Keywords: writer's cram; musician dystonia; TMS; zolpidem
MeSH Terms: conditions — Dystonic Disorders | interventions — Zolpidem

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Patients with focal dystonia treatment first placebo second (Active Comparator): Zolpidem 5 mg single dose
  Interventions: Drug: Zolpidem
- Patients with focal dystonia placebo first treatment second (Placebo Comparator): Placebo 5 mg single dose
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Zolpidem — Patients will undergo transcranial magnetic stimulation, 18F-FDG-PET brain imaging, and clinical testing after a single 5 mg dose of Zolpidem.
  Arms: Patients with focal dystonia treatment first placebo second
Drug: Placebo — Patients will undergo transcranial magnetic stimulation, 18F-FDG-PET brain imaging, and clinical testing after a single dose of placebo.
  Arms: Patients with focal dystonia placebo first treatment second

SUMMARY:
To study electrophysiological and imaging correlations of the clinical effectiveness of zolpidem in task-specific dystonia and to elucidate mechanisms underlying its therapeutic effects, patients with focal dystonia will be clinically evaluated and will undergo transcranial magnetic stimulation and FDG-PET CT brain imaging after a single 5 mg dose of zolpidem and placebo, in two separate sessions. Resting motor threshold (RMT), active motor threshold (AMT), resting and active input/output (IO) curve, short-interval intracortical inhibition (SICI) curve, long interval intracortical inhibition (LICI), intracortical facilitation (ICF), and cortical silent period (CSP) will be measured. Objective clinical improvement will be rated using Burke-Fahn-Marsden Dystonia Rating Scale-movement (BFM-M) and writer's cramp rating scale (WCRS). Subjective improvement will be measured using the visual analog scale (VAS). Only a subset of patients (10 patients) will undergo positron emission tomography with 18F-2-fluoro-2-deoxy-D-glucose (18F-FDG PET) brain imaging after a single 5 mg dose of zolpidem and placebo.

DETAILED DESCRIPTION:
Background: The present view of dystonia is as of a circuit disorder, involving basal ganglia-thalamo-cortical and cerebello-thalamo-cortical pathways. One of the key pathophysiological features of dystonia is decreased inhibition at several levels of the central nervous system. The lack of inhibition may account for many of the dystonic symptoms, such as co-contraction of antagonistic muscles, loss of selectivity in muscle activation during movement, or overflow of dystonic symptoms in body parts not engaged in the movement. Gamma-aminobutyric acid (GABA) is the main inhibitory neurotransmitter in the central nervous system (CNS). Studies in animal models, as well as neuroimaging and electrophysiological data on dystonic patients, provide evidence of abnormal GABA neurotransmission in dystonia. Currently, there is no cure for dystonia, but there are several symptomatic treatment options, including medications and surgical approaches. While only a minority of dystonia patients is eligible for deep brain stimulation most affected individuals are dependent on pharmacological treatments for symptomatic relief. These include botulinum toxin injections and oral medications. Botulinum toxin injection treatment is effective in focal and segmental dystonia, but it requires repeated injections, may be associated with resistance to treatment, and is expensive. Available oral medications are however not very effective (particularly in adult dystonia patients) and may be associated with intolerable adverse effects. Consequently, research into the use of new pharmaceuticals approaches is warranted. Zolpidem is a widely used hypnotic agent that potentiates GABA transmission, as a selective agonist of the benzodiazepine subtype receptor α1. Zolpidem has been recently reported in an open-labeled study to be effective in primary focal and generalized dystonia, with the effect being variable among different dystonia patients.

Aims: To study electrophysiological correlations of the clinical effectiveness of zolpidem in task-specific dystonia and to elucidate mechanisms underlying its therapeutic effects, which have not yet been investigated.

Hypotheses: Taking into account reports in the literature, we believe we will be able to prove zolpidem is more effective in improving focal dystonia than placebo. Since zolpidem acts as an agonist in GABA-A receptors, we believe it will enhance TMS measures that are known to be mediated true GABA-A signaling. We hypothesize that the effects of zolpidem on electrophysiological measures will correlate with the patient's response to treatment.

Patients and inclusion/exclusion criteria: Thirty patients with writer's cramp or musician dystonia will be recruited from the outpatient clinic for extrapyramidal disorders. Patients treated with botulinum toxin within the last 3 months and patients with contraindications for TMS will be excluded. Patients will not be allowed to take benzodiazepines, zolpidem, or other sedative drugs for 48 hours prior to the experiment. No changes in medications before and during the whole study apart from study-related drug intervention will be allowed.

Study protocol: 30 patients will undergo TMS after a single 5 mg dose of zolpidem and placebo, in two separate sessions. Objective clinical improvement will be rated using Burke-Fahn-Marsden Dystonia Rating Scale-movement (BFM-M) and writer's cramp rating scale (WCRS). Subjective improvement will be measured using the visual analog scale (VAS). In addition, 10 patients will undergo positron emission tomography with 18F-2-fluoro-2-deoxy-D-glucose (18F-FDG PET) brain imaging after a single 5 mg dose of zolpidem and placebo.

Methods:

Transcranial magnetic stimulation (TMS) Single TMS pulses will be applied using Magstim 2002 magnetic stimulator with monophasic waveform (Magstim Company, Carmarthenshire, Wales, UK). For double TMS pulses, we will use two Magstim 2002 stimulators connected with the Bistim module. The stimulators will be connected to a standard figure 8 coil. The coil will be positioned tangentially to the skull and over the 'hotspot' point on the scalp, with the handle pointing backward at an angle of ~ 45 ° with respect to the sagittal plane. Hotspot point is defined as stimulation site resulting in the largest motor evoked potentials (MEPs) recorded over the contralateral abductor pollicis brevis (APB) muscle. A hotspot point will be found by visual inspection. The MEP amplitude in APB muscle will be measured with electromyography (EMG).

Statistical analysis: Clinical and TMS measures on zolpidem and placebo will be compared using parametric or nonparametric T-test or repeated-measures ANOVA. Correlations will be tested using Spearman analysis. Statistical parametric mapping (SPM8; paired t-test, p<0.001) will be used to identify the zolpidem effect on global brain metabolism.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of writer's cramp or musician dystonia

Exclusion Criteria:

* Patients treated with botulinum toxin within the last 3 months
* Patients with contraindications for TMS
* Patients taking benzodiazepines, zolpidem or other sedative drugs 48 hours prior to the experiment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2017-09-30 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Change in the transcranial magnetic stimulation measures between zolpidem 5 mg and placebo | 30 minutes after the intervention
  Transcranial magnetic stimulation measures (resting and active cortical motor threshold, resting and active input-output curve, short intracortical inhibition, long intracortical inhibition, intracortical facilitation) after zolpidem 5 mg and placebo will be compared.
Change in brain metabolism detected on FDG-PET CT brain imaging between zolpidem 5 mg and placebo | 30 minutes after the intervention
  FDG-PET CT brain imaging

SECONDARY OUTCOMES:
Change in The Burke-Fahn-Marsden Dystonia Rating Scale (BFMS) between zolpidem 5 mg and placebo | 30 minutes after the intervention
  Dystonia can be objectively assessed using the BFMS. The BFMS is subdivided into a movement scale and a disability scale. Only the movement scale will be used. The minimum total score is 0, the maximal total score is 120. Patients who are more affected with dystonia get higher scores.

OTHER OUTCOMES:
Change in The Writer's Cramp Rating Scale (WCRS) between zolpidem 5 mg and placebo | 30 minutes after the intervention
  The writer's cramp dystonia can be objectively assessed using WCRS. The minimum score on WCRS is 0 and the maximum score is 30. The WCRS consists of two subscores, the writing movement score with the minimum score 0 and the maximum score 28 and the writing speed score with the minimum score 0 and the maximum score 2. The higher the score, the more is a patient affected with the writer's cramp dystonia.
Change in the Visual Analog Score between zolpidem 5 mg and placebo | 30 minutes after the intervention
  To subjectively assess dystonia, the Visual Analog Scale will be used. The minimum score on the scale will be 0 and the maximum score will be 10. A higher score will mean a greater impairment due to the presence of dystonia.

CONTACTS AND LOCATIONS:
Overall Officials: Maja Kojović, PhD, MD, Principal Investigator — University Medical Centre Ljubljana
Locations (2):
- University Clinical Centre of Serbia, Belgrade, Serbia
- Departmet of Neurology, University Medical Centre Ljubljana, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: No
If I will be contacted by other researchers after publication I will share individual participant data that will underlie published results.

REFERENCES:
- [Background] Lehericy S, Tijssen MA, Vidailhet M, Kaji R, Meunier S. The anatomical basis of dystonia: current view using neuroimaging. Mov Disord. 2013 Jun 15;28(7):944-57. doi: 10.1002/mds.25527. PMID 23893451
- [Background] Kapogiannis D, Wassermann EM. Transcranial magnetic stimulation in Clinical Pharmacology. Cent Nerv Syst Agents Med Chem. 2008 Dec;8(4):234-240. doi: 10.2174/187152408786848076. PMID 19122782
- [Background] Quartarone A, Hallett M. Emerging concepts in the physiological basis of dystonia. Mov Disord. 2013 Jun 15;28(7):958-67. doi: 10.1002/mds.25532. PMID 23893452
- [Background] Thenganatt MA, Jankovic J. Treatment of dystonia. Neurotherapeutics. 2014 Jan;11(1):139-52. doi: 10.1007/s13311-013-0231-4. PMID 24142590